CLINICAL TRIAL: NCT02731027
Title: Biomarkers of Spontaneous Recovery From Traumatic Spinal Cord Injury
Acronym: SCIMARK
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); New York State Department of Health (Other Government); University of Louisville (Other); Kessler Foundation (Other); Thomas Jefferson University (Other); University of British Columbia (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Ona Bloom, Principal Investigator, Northwell Health
Other Study IDs: 14612
Record Dates: First submitted 2016-03-17; First posted 2016-04-07 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls
- Participants with Spinal Cord Injury

SUMMARY:
The purpose of the study is to profile biochemical responses and measure functional recovery in parallel, throughout the 1st year after spinal cord injury (SCI), within the same participants. These responses and recovery will be evaluated in samples from people who have had a spinal cord injury due to trauma (e.g. car accident or a fall) within the first year after SCI. Specifically, the investigators will test the hypothesis that a subset of inflammatory biomarkers correlate inversely with functional recovery. The investigators will use these data to build a predictive model of functional recovery after SCI that incorporates biomarkers that can be easily quantified in the clinic.

Total anticipated enrollment will be 100 participants with SCI across three different sites (Northwell Health System (NY), The Kessler Institute for Rehabilitation (NJ), University of Louisville (KY) and may enroll up to 30 participants without SCI.

DETAILED DESCRIPTION:
At all study visits, a member of the study team (investigator) will collect basic demographic and health information from the participant or the participant's medical record.

Study participants will have blood drawn at each study visit (approximately 2 tablespoons). The participant will be asked to partake in 4 study visits over the course of 1 year. The first visit will be within the first 0-14 days of SCI. The 2nd, 3rd, and 4th visits will be 3, 6, and 12 months after their spinal cord injury.

At study visits 2, 3 and 4, a study investigator will also perform some clinical evaluations for research purposes to test how the participant is recovering the ability to perform activities of daily living and move after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

SCI Subject Inclusion Criteria: To be eligible for prospective enrollment, participants are required to meet the following inclusion criteria:

* ≥18 years old with traumatic SCI
* Injury within 0-3 days post injury prior to enrollment
* All American Spinal Injury Association (ASIA) grade classification A-D.
* Neurological injury level C4-T10

Exclusion Criteria:

To be eligible for prospective enrollment, SCI subjects are required to not meet the following exclusion criteria:

* Stage III-IV pressure ulcers
* Cancer, chemotherapy, neutropenia
* Pregnancy (all female trauma patients of childbearing years are given a pregnancy test on admission as part of routine admitting labs) or lactation
* No known previous SCI
* Autoimmune disease
* Pre-existing neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will conduct an observational, prospective, longitudinal, multi-site study of traumatic SCI patients within 0-3 days of the initial injury and throughout the first year post SCI.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-10; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Circulating inflammatory response from the peripheral blood for each SCI participant | 1 year
  Sample 1 will take place at the earliest possible time within 0-3 days post SCI. All blood products will be collected with strict adherence to universal precautions, and whenever possible, will occur concurrently with clinical blood draws. Blood samples collected from patients with documented concurrent infections such as UTI, as indicated by fever, hematuria or increased spasticity with the presence of pyuria (>25 wbc/high power field), which will raise inflammatory biomarker levels independent of SCI, will be analyzed as a subgroup.
ASIA Impairment Scale (AIS) Grade for each SCI participant | 1 year
  The AIS grade will be the primary functional outcome measure. Data will be collected once acutely (0-3 days), and at 3, 6, and 12 months after SCI.

SECONDARY OUTCOMES:
Spinal Cord Independence Measure (SCIM) for each SCI participant | 1 year
  The SCIM score will be a secondary measure to assess sensitivity to changes in ability to perform activities of daily living and facilitate a multiscale correlative analysis with biochemical variables measured. Data will be collected once at 3, 6, 12 months after SCI.
Neuromuscular Recovery Scale (NRS) for each SCI participant | 1 year
  To assess ability to perform tasks related to mobility, standing and walking for each SCI participant. Data will be collected once at 3,6,12 months after SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Ona Bloom, Ph.D., Principal Investigator — Northwell Health System
Locations (6):
- United States (5):
  - Frazier Rehab Institute, Univ. of Louisville, Louisville, Kentucky
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - The Feinstein Institute for Medical Research, Northwell Health, Manhasset, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No